CLINICAL TRIAL: NCT00947661
Title: Efficacy and Safety of SPARC0912 and Reference0912 in Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLR_09_12
Record Dates: First submitted 2009-07-23; First posted 2009-07-28 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: glaucoma latanoprost
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- SPARC0912 (Experimental): Test drug
  Interventions: Drug: SPARC0912
- Reference0912 (Experimental): Reference drug
  Interventions: Drug: Reference0912

INTERVENTIONS:
Drug: SPARC0912 — Eye drops, once daily, 12 weeks
  Arms: SPARC0912
Drug: Reference0912 — Eye drops, once daily, 12 weeks
  Arms: Reference0912

SUMMARY:
A single-blind , 12-week, parallel group clinical study is planned to evaluate the efficacy and safety of SPARC0912 and Reference0912. SPARC0912 is an experimental drug having similar active ingredient but containing a different preservative as that in Reference0912. Patients with open angle glaucoma or ocular hypertension will be enrolled and randomly assigned to receive either product. One drop will be instilled to the study eye nightly at 8:00 PM.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years.
* Diagnosis of ocular hypertension (OHT) or primary open angle glaucoma (POAG).
* Unmedicated IOP ≥ 22 mmHg in one or both eyes.
* Given informed consent.
* Women of child bearing potential practicing an acceptable method of birth control with a negative urine pregnancy test.

Exclusion Criteria:

* Known lack of ocular hypotensive response to topical ophthalmic, prostaglandin analogs (in the opinion of the investigator).
* Intraocular conventional surgery or laser surgery within the past six months.
* Refractive surgery in study eye (e.g., radial keratotomy, PRK, LASIK, etc.) within the past 3 months.
* Angle closure glaucoma or a history of acute angle closure treated with a peripheral iridotomy.
* Ocular trauma within the past 3 months.
* Progressive retinal or optic nerve disease apart from glaucoma.
* Concurrent infectious/non infectious conjunctivitis, keratitis, or uveitis in either eye.
* Any abnormality preventing stable applanation tonometry.
* Use of contact lens for the duration of the study.
* Any opacity or subject uncooperativeness that restricts adequate examination of the ocular fundus or anterior chamber.
* Clinically significant ocular disease (e.g., corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications is not judged safe.
* Clinically significant systemic disease which might interfere with the study.
* History of non-compliance to medical regimens or unwilling to comply with the study protocol.
* Participation in another clinical study within the last thirty (30) days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC study site, High Point, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SPARC0912: SPARC0912 administered once daily for 12 weeks
- Reference0912: Reference0912 administered once daily for 12 weeks
Period: Overall Study
Arm/Group | SPARC0912 | Reference0912
Started | 289 | 289
Completed | 276 | 274
Not Completed | 13 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPARC0912 | Reference0912 | Total
Number analyzed (Participants) | 289 | 289 | 578
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (9.59) | 63.8 (11.08) | 63.4 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 188 | 374
  Male | 103 | 101 | 204

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure From Baseline to Week 12
Description: 95% CI for the difference between treatment groups in estimated mean change from baseline was computed for each a total of 12 time points (for the reduction in intraocular pressure from baseline to Week 12)
Time Frame: 12 weeks
Population: Intent to treat population without LOCF
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- SPARC0912: The change from baseline in intraocular pressure was calculated. A positive change from baseline suggested a reduction from baseline in intraocular pressure. Change from baseline was analyzed using an analysis of covariance methodology, a two-sided 95% CI for the difference between treatment groups in estimated mean change from baseline (i.e., LS means derived from the ANCOVA model) was computed for each time point at each visit (a total of 12 time points at 4 visits i.e. 3 time points at each visit).
Arm/Group | SPARC0912 | Reference0912
Number analyzed (Participants) | 275 | 276
mm Hg | 6.12 (0.23) | 6.91 (0.23)
Statistical Analysis 1: Comparison: SPARC0912; Test type: Non-Inferiority or Equivalence — Analysis of covariance included treatment, site, and intraocular pressure group as a covariate. Two-sided 95% confidence interval for the difference between treatment groups in estimated mean change from baseline lease square means was computed for each time point. Non-inferiority of SPARC drug relative to Reference was established if: 95% confidence interval included 0, the upper limit of the 95% CI was <1.5, and upper limit of 95% CI was <1 at most (at least 7 of 12) time point; p < 0.01, ANCOVA

ADVERSE EVENTS:
Groups:
- SPARC0912: SPARC's formulation administered once daily for 12 weeks
- Reference0912: Reference formulation administered once daily for 12 weeks
Arm/Group | SPARC0912 | Reference0912
Serious Adverse Events (participants affected / at risk) | 3/289 | 5/289
Other Adverse Events (participants affected / at risk) | 3/289 | 4/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPARC0912 (N=289) | Reference0912 (N=289)
Macular edema (Eye disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Colitis (General disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Elevated blood pressure (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPARC0912 (N=289) | Reference0912 (N=289)
abdominal pain, colitis (Gastrointestinal disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Back pain, Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other